CLINICAL TRIAL: NCT02675140
Title: Chengdu Women's and Children's Central Hospital
Brief Title: Effect of Hookworm Elimination and Vitamin A Intervention on Iron Status of Preschool Children in Sichuan, China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chengdu Maternal and Children's Health Care Hospital (Other)
Responsible Party: Principal Investigator, Ke Chen, chief, Chengdu Maternal and Children's Health Care Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChengduWCCH
Record Dates: First submitted 2015-08-28; First posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Anemia; Worm Infections
MeSH Terms: conditions — Anemia; Helminthiasis | interventions — Albendazole; Vitamin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ZENTEL (Experimental): Children in intervention group 1 was received 400 mg single-dose albendazole administration, by mouth, for once.
  Interventions: Drug: ZENTEL
- ZENTEL and Vitamin A Soft Capsules (Experimental): Children in intervention group 2 was received a 200,000 IU vitamin A capsule combined 400 mg single-dose albendazole once initially, by mouth.
  Interventions: Drug: ZENTEL and Vitamin A Soft Capsules
- No drug adminitrated (No Intervention): Children in this Group were received no intervention as control group

INTERVENTIONS:
Drug: ZENTEL — Children in Group 2 (n=62) received 400 mg single-dose albendazole (helmintic treatment)
  Other Names: albendazole
  Arms: ZENTEL
Drug: ZENTEL and Vitamin A Soft Capsules — Children in Group 3 (n=60) received a 200,000 IU vitamin A capsule combined with 400 mg single-dose albendazole once initially
  Other Names: albendazole and vitamin A
  Arms: ZENTEL and Vitamin A Soft Capsules

SUMMARY:
The present study is intended to supplement the preschool anemic children with vitamin A capsule and de-hookworm administration in poverty Sichuan province. We eventually expect our study can provide a cost-effective, safe and more beneficial public health strategy to manage the anemia status of preschool children in poverty area.

DETAILED DESCRIPTION:
Subjects and ethical approval This randomized, control and double-blinded cohort study was performed in Dayi, Pixian and Meishan country, Sichuan Province, western China, which are suburbs of Chengdu city with a low class of socioeconomic status, from March 2012 to September 2014 and approximately about 216 anemic preschool children aged 3-6 years were randomly recruited from nine kindergartens of the three countries for the study during intervention period. The eligibility criteria for participation were as follows: 1) apparent health; 2) Hb concentration <110 g/l but not <80 g/l; 3) C-reaction protein (CRP) <10 mg/L; 4) parental or guardian approval of participation in all aspects of the study; and 5) parental/guardian agreement to avoid the additional use of vitamin and mineral supplements and de-hookworm administration during the trial. Children with Hb<80 g/l and /or CRP >10 mg/l were sent to hospital with special treatment.

We conducted a census in each regional kindergarten to determine which households included an eligibility preschool children. Then field health workers conducted a family survey to determine which children was included. Eligible families were visited by a field worker who explained the protocol, answered questions, and obtained written informed consent from parents/guardians. The enrollment and research plan were reviewed and approved by the institutional ethics committee of the Chengdu Women's and Children's Central Hospital of Chongqing Medical University in Sichuan province, China. The present study complied with the code of ethics of the World Medical Association (Declaration of Helsinki).

The primary objective for the present study was to measure the change in serum Hb before and after intervention. A sample size of about 60 anemic preschool children per group was required to detect an absolute difference of 10 g/L of Hb concentration among three intervention groups after supplementation with 95% power and α= 0.05 for a two-sided two-sample t-test. To allow for 20% rate of dropout over the duration of the study, we initially planed to recruit about 72 anemic children per group (totally 216). We estimated that the prevalence of anemia of preschool children in locality was about 16%[17], eventually about 1350 children were recruited into an initial Hb screening study before intervention and about 450 for each group.

Intervention All eligible anemic children were randomly divided into three groups: Group 1 was received no intervention as control group; Group 2 was received 400 mg single-dose albendazole administration and Group 3 was received a 200,000 IU vitamin A capsule combined 400 mg single-dose albendazole once initially. For ethical reason, all of the children in control group were given a single-dose albendazole at the end of study. Immediately after recruitment, children in one class were assigned a study number that had been previously randomly assigned to the intervention or control group with fixed, equal allocation to each group prepared by a third party. The RAND function of Excel (Microsoft, Redmond, WA, USA) was used to generate computer randomly permutated codes. The physicians, nurses, field health workers, parents, children and laboratory personnel were blinded to the treatment assignment of each child throughout the study period. The data manager, statistician, and all investigators remained blinded to group assignments until the end of data analysis. The total duration of intervention and evaluation were six months. Vitamin A capsule and albendazole tablet were provided by Sichuan Pearl Pharmaceutical Co., Ltd.

Compliance Compliance of albendazole tablet and vitamin A capsule were monitored using recording tables, in which teachers recorded whether the child consumed "all" or "none" of the albendazole tablet and vitamin A capsule. To avoid exchange of albendazole tablet and vitamin A capsule by classmates, the three groups were physically separated by being moved to opposite corners of the classroom. Distribution and consumption of the albendazole tablet and vitamin A capsule took place under close supervision; children in group 2 and group 3 were not allowed to leave the classroom or return to their original seats before they had finished eating their albendazole tablet and vitamin A capsule. The distribution of tablets was performed by nursery managers, but not health care workers and nursery teachers. Information on the acceptability of the albendazole tablet and vitamin A capsule was obtained by a short questionnaire after administered.

Questionnaire interview A 30-minute questionnaire was conducted by a trained interviewer after recruitment. The questionnaire included questions on demographic information (children's age, sex), educational levels of main caregivers ( who were at least responsible for the half of care time of children), monthly family income, use of vitamin/mineral supplement before trial and food frequency recall (the frequency of deep-colored vegetables and milk, liver and egg).

Anthropometric measurements Anthropometric examinations were conducted by the same trained anthropometric nurse at baseline and follow-up (6-mo) time points using standardized techniques to eliminate intra-examiner error. Duplicate measurements were performed for all children. The inter-examiner coefficient of variation of weight and height for each examiner in each group was less than 5%. Weight was recorded using a weighing scale (100Med, Beijing, China) to the nearest 100 g with subjects in minimal clothing and bare feet. Similarly, height was measured in the standard position by a height scale (Haode, Guangzhou, China) to the nearest 0.1 cm. By using reference data from World Health Organization (WHO; 2005), the Z-scores were calculated for height for age (HAZ), weight for height (WHZ), and weight for age (WAZ). All indices were computed using Anthro (2005) for the personal computer, as recommended by the WHO (http://www.who.int/childgrowth/software/en/).

Blood sample collection and biochemical assessment At the beginning and at 3 and 6 month after intervention, three blood samples (about 1 mL) were collected by venipuncture of an antecubital vein from each subject before breakfast in hospital. A quarter of a milliliter was drawn into a container containing heparin to measure Hb by the hemoglobincyanide method (Maker, Chengdu, China). The interassay variation was lower than 5% and the intra-assay variation was lower than 10%. The blood samples were immediately stored at 4° C to prevent micro-hemolysis and were separated within 5 h. The remaining blood was centrifuged at 3000g for 5 min at room temperature. The centrifuged serum samples were divided into aliquots and immediately transported to the laboratory and stored at -20°C. The concentrations of serum ferritin (SF) were measured using a commercial enzyme-linked immunosorbent assay (ELISA) (Sunbiote, Shanghai, China). Serum soluble transferrin receptor (sTfR) was measured by microparticle-enhanced immunoassay (Sunbiote, Shanghai, China). CRP was measured by particle-enhanced immunoturbidimetry (Sunbiote, Shanghai, China). Serum retinol concentration was determined by using high-performance liquid chromatography. Serum retinol was measured by experienced examiners in the Pediatric Laboratory of Chongqing Medical University and the other biochemical indices in Clinical Laboratory Center of Chengdu Women & Children's Central Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Apparent health
2. Hb concentration <110 g/l but not <80 g/l
3. C-reaction protein (CRP) <10 mg/L
4. Parental or guardian approval of participation in all aspects of the study
5. Parental/guardian agreement to avoid the additional use of vitamin and mineral supplements and de-hookworm administration during the trial.-

Exclusion Criteria:

1) Children with Hb<80 g/l and /or CRP >10 mg/l were sent to hospital with special treatment

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 209 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Hemoglobin concentration | six month

IPD SHARING:
Plan to Share IPD: Yes
It is my pleasure to share some data with other researcher who are interested in this theme.